CLINICAL TRIAL: NCT00291343
Title: Booster Vaccination Study to Assess Immunogenicity & Safety of a Dose of GSK Biologicals' Mencevax™ ACWY & 1/5th of a Dose of Mencevax™ ACWY in Subjects Primed in the DTPW-HBV=HIB-MENAC-TT-011 Study
Brief Title: Immune Response & Safety of GSK Biologicals' Mencevax™ ACWY in Subjects Primed in the DTPW-HBV=HIB-MENAC-TT-011 Study
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 105239 (mth24-30); 105245 (Other: GSK)
Record Dates: First submitted 2006-02-13; First posted 2006-02-14 (Estimated); Results first posted 2017-08-03 (Actual); Last update posted 2018-06-06 (Actual); Status verified 2017-04

CONDITIONS: Infections, Meningococcal
Keywords: hepatitis B; meningococcal vaccine; pertussis; Prophylaxis diphtheria; meningococcal serogroups A and C diseases; tetanus; Haemophilus influenzae type b
MeSH Terms: conditions — Meningococcal Infections; Hepatitis B; Whooping Cough; Tetanus; Haemophilus Infections | interventions — Hiberix

ARMS (2):
- TRITANRIX™-HEPB/HIB-MENAC +MENCEVAX™ ACWY GROUP (Experimental): Subjects previously primed with 3 doses of Tritanrix™-HepB/Hib-MenAC vaccine in study NCT00290303, were administered in the current study one booster dose of Tritanrix™-HepB/Hiberix™, intramuscularly in the left anterolateral thigh, at 15-24 months of age and one booster dose of Mencevax™ ACWY by subcutaneous injection in the upper region of the left arm, at 24-30 months of age.
  Interventions: Biological: Tritanrix™- HepB; Biological: Hiberix™; Biological: Mencevax™ ACWY
- TRITANRIX™-HEPB/HIBERIX™+MENCEVAX™ ACWY GROUP (Active Comparator): Subjects previously primed with 3 doses Tritanrix™-HepB/Hiberix™ vaccine in study NCT00290303, were administered in the current study one booster dose of Tritanrix™-HepB/Hiberix™, intramuscularly in the left anterolateral thigh, at 15-24 months of age and one dose of Mencevax™ ACWY by subcutaneous injection in the upper region of the left arm, at 24-30 months of age.
  Interventions: Biological: Tritanrix™- HepB; Biological: Hiberix™; Biological: Mencevax™ ACWY

INTERVENTIONS:
Biological: Tritanrix™- HepB — One intramuscular dose during the booster vaccination study in subjects aged 15 to 24 months
Biological: Hiberix™ — One intramuscular dose during the booster vaccination study in subjects aged 15 to 24 months
Biological: Mencevax™ ACWY — One full subcutaneous dose in subjects aged 24 to 30 months or 1/5th of a dose intramuscular in subjects aged 30 to 36 months

SUMMARY:
This study will be conducted in three stages. In the DTP booster stage at 15 to 24 months of age, all subjects will receive a booster dose of Tritanrix™-HepB/Hiberix™. In the Mencevax™ ACWY "full dose" stage at 24 to 30 months of age all subjects will receive a dose of Mencevax™ ACWY. In the Mencevax™ ACWY "small dose" stage at 30 to 36 months of age, the first 75 subjects in each of the two centers will be tested for boostability of the MenA and MenC immune response by giving a fifth of a dose of a Mencevax™ ACWY vaccine. The Protocol Posting has been updated in order to comply with the FDA Amendment Act, Sep 2007.

DETAILED DESCRIPTION:
Subjects in the group that was previously primed with Tritanrix™-HepB/Hiberix™ will be the control group for the group that was previously primed with Tritanrix™-HepB/Hib-MenAC.

Blood samples will be drawn from subjects as follows:

* prior to and one month after the full dose of the Mencevax™ ACWY vaccine.
* prior to and one month after 1/5th of a dose of Mencevax™ ACWY vaccine (only for the first 75 subjects in each of the two centers).

ELIGIBILITY:
Inclusion criteria:

* Subjects who the investigator believes that their parents/guardians can and will comply with the requirements of the protocol.
* A male or female between, and including, 15 and 24 months of age at the time of vaccination.
* Written informed consent obtained from the parent or guardian of the subject.
* Healthy subjects as established by medical history and clinical examination before entering into the study.
* Having participated in the primary vaccination study DTPW-HBV=HIB-MENAC-TT-011 (eTrack No. 100478) in Center No. 4328 or Center No.4329.

Exclusion criteria:

* Use of any investigational or non-registered product (drug or vaccine) other than the study vaccine within 30 days preceding the vaccination, or planned use during the study period.
* Chronic administration (defined as more than 14 days) of immunosuppressants or other immune-modifying drugs within six months prior to vaccination.
* Planned administration/ administration of a vaccine not foreseen by the study protocol within 30 days of vaccination; with the exception of oral poliovirus vaccine (OPV).
* Booster vaccination against diphtheria, tetanus, pertussis, hepatitis B, Haemophilus influenzae type b (Hib) and/or meningococcal serogroups A and/or C disease, after the date of the study conclusion visit of the primary vaccination study DTPW-HBV=HIB-MENAC-TT-011 (eTrack No. 100478).
* History of diphtheria, tetanus, pertussis, hepatitis B, Hib and/or meningococcal serogroup A or C disease.
* Known exposure to diphtheria, tetanus, pertussis, hepatitis B, Hib and/or meningococcal serogroup A or C disease.
* Any confirmed or suspected immunosuppressive or immunodeficient condition, based on medical history and physical examination.
* A family history of congenital or hereditary immunodeficiency.
* History of allergic disease or reactions likely to be exacerbated by any component of the vaccine.
* Major congenital defects or serious chronic illness.
* History of any neurologic disorders or seizures including febrile seizures in infancy.
* Acute disease at the time of enrolment.
* Planned or actual administration of immunoglobulins and/or any blood products within the three months preceding Mencevax™ ACWY vaccination.

Ages: 15 Months to 24 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 296 (Actual)
Dates: Start 2006-02-01; Primary Completion 2007-03-15 (Actual); Study Completion 2007-03-15 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (2):
- Philippines (2):
  - GSK Investigational Site, Manila
  - GSK Investigational Site, Sampaloc, Manila

IPD SHARING:
Plan to Share IPD: Yes
Patient-level data for this study will be made available through www.clinicalstudydatarequest.com following the timelines and process described on this site.

REFERENCES:
- See also: Researchers can use this site to request access to anonymised patient level data and/or supporting documents from clinical studies to conduct further research. — https://www.clinicalstudydatarequest.com
- Available data/document: Study Protocol: 105239 (mth24-30) — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Informed Consent Form: 105239 (mth24-30) — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Dataset Specification: 105239 (mth24-30) — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Clinical Study Report: 105239 (mth24-30) — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Individual Participant Data Set: 105239 (mth24-30) — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register. The results of this study 105239 are summarised with study 105245 on the GSK Clinical Study Register.
- Available data/document: Statistical Analysis Plan: 105239 (mth24-30) — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register

RESULTS

PARTICIPANT FLOW:
Groups:
- Tritanrix-HepB/Hib-MenAC +Mencevax ACWY Group: Subjects previously primed with 3 doses of Tritanrix-HepB/Hib-MenAC vaccine in study NCT00290303, were administered in the current study one booster dose of Tritanrix-HepB/Hiberix, intramuscularly in the left anterolateral thigh, at 15-24 months of age and one booster dose of Mencevax ACWY by subcutaneous injection in the upper region of the left arm, at 24-30 months of age.
- Tritanrix-HepB/Hiberix+Mencevax ACWY Group: Subjects previously primed with 3 doses Tritanrix-HepB/Hiberix vaccine in study NCT00290303, were administered in the current study one booster dose of Tritanrix-HepB/Hiberix, intramuscularly in the left anterolateral thigh, at 15-24 months of age and one dose of Mencevax ACWY by subcutaneous injection in the upper region of the left arm, at 24-30 months of age.
Period: Overall Study
Arm/Group | Tritanrix-HepB/Hib-MenAC +Mencevax ACWY Group | Tritanrix-HepB/Hiberix+Mencevax ACWY Group
Started | 203 | 93
Completed | 203 | 93
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Tritanrix-HepB/Hib-MenAC +Mencevax ACWY Group | Tritanrix-HepB/Hiberix+Mencevax ACWY Group | Total
Number analyzed (Participants) | 203 | 93 | 296
Age, Continuous [Mean (Standard Deviation); unit: Months] | 24.2 (0.68) | 24.1 (0.40) | 24.17 (0.61)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 94 | 42 | 136
  Male | 109 | 51 | 160

OUTCOME MEASURES:

1. Primary Outcome: Number of Subjects With Serum Bactericidal Activity Against Neisseria Meningitidis Serogroups A, C (rSBA-MenA, C) Using Rabbit Complement Antibodies
Description: Antibody cut-offs were higher than or equal to (≥) 1:128
Time Frame: 1 month after Mencevax ACWY vaccination (at 25 to 31 months of age).
Population: The analyses were performed on the Booster ATP cohort for immunogenicity which included all subjects who had received 3 doses in the primary vaccination study, who had received a single dose of MenACWY according to protocol at 24 to 30 months of age and for whom data concerning immunogenicity measures were available.
Measure: Number; unit: Subjects
Arm/Group | Tritanrix-HepB/Hib-MenAC +Mencevax ACWY Group | Tritanrix-HepB/Hiberix+Mencevax ACWY Group
Number analyzed (Participants) | 192 | 67
Subjects
  rSBA-MenA ≥1:128: number analyzed (Participants) | 116 | 66
  rSBA-MenA ≥1:128 | 116 | 66
  rSBA-MenC ≥1:128 | 192 | 53

2. Secondary Outcome: Number of Subjects With Anti-rSBA-MenA, C Antibody Titers ≥ Pre-defined Cut-off Values
Description: Pre-defined cut-offs were ≥ 1:8 and ≥ 1:128
Time Frame: Prior to (at 24 to 30 months of age) and after (at 25 to 31 months of age) Mencevax ACWY vaccination.
Population: The analysis were performed on the Booster ATP cohort for immunogenicity which included all subjects who had received 3 doses in the primary vaccination study, who had received a single dose of MenACWY according to protocol at 24 to 30 months of age and for whom data concerning immunogenicity measures were available.
Measure: Number; unit: Subjects
Arm/Group | Tritanrix-HepB/Hib-MenAC +Mencevax ACWY Group | Tritanrix-HepB/Hiberix+Mencevax ACWY Group
Number analyzed (Participants) | 192 | 67
Subjects
  rSBA-MenA ≥1:8 (M24-30): number analyzed (Participants) | 169 | 60
  rSBA-MenA ≥1:8 (M24-30) | 164 | 56
  rSBA-MenA ≥1:8 (M25-31): number analyzed (Participants) | 116 | 66
  rSBA-MenA ≥1:8 (M25-31) | 116 | 66
  rSBA-MenA ≥1:128 (M24-30): number analyzed (Participants) | 169 | 60
  rSBA-MenA ≥1:128 (M24-30) | 157 | 55
  rSBA-MenC ≥1:8 (M24-30): number analyzed (Participants) | 180 | 63
  rSBA-MenC ≥1:8 (M24-30) | 166 | 22
  rSBA-MenC ≥1:8 (M25-31) | 192 | 61
  rSBA-MenC ≥1:128 (M24-30): number analyzed (Participants) | 180 | 63
  rSBA-MenC ≥1:128 (M24-30) | 98 | 16

3. Secondary Outcome: Anti-rSBA-MenA, C Antibody Titers
Description: Antibody titers were expressed as Geometric Mean Titers (GMTs)
Time Frame: Prior to (at 24 to 30 months of age) and after (at 25 to 31 months of age) Mencevax ACWY vaccination.
Population: as for outcome 2
Measure: Geometric Mean (95% Confidence Interval); unit: Titers
Arm/Group | Tritanrix-HepB/Hib-MenAC +Mencevax ACWY Group | Tritanrix-HepB/Hiberix+Mencevax ACWY Group
Number analyzed (Participants) | 192 | 67
Titers
  rSBA-MenA (M24-30): number analyzed (Participants) | 169 | 60
  rSBA-MenA (M24-30) | 551.9 [459.6 to 662.6] | 469.1 [320.3 to 687.0]
  rSBA-MenA (M25-31): number analyzed (Participants) | 116 | 66
  rSBA-MenA (M25-31) | 2018.9 [1778.0 to 2292.3] | 2108.1 [1733.4 to 2563.9]
  rSBA-MenC (M24-30): number analyzed (Participants) | 180 | 63
  rSBA-MenC (M24-30) | 120.6 [99.3 to 146.5] | 15.5 [9.4 to 25.6]
  rSBA-MenC (M25-31) | 11024.4 [9394.5 to 12937.0] | 437.2 [269.6 to 708.9]

4. Secondary Outcome: Number of Subjects With Anti-pilysaccharide A and C (Anti-PSA/PSC) Antibody Concentrations ≥ Predefined Cut-off Values
Description: Antibody cut-offs were ≥ 0.3, 2 micrograms per millilitre (µg/mL).
Time Frame: Prior to (at 24 to 30 months of age) and after (at 25 to 31 months of age) Mencevax ACWY vaccination.
Population: as for outcome 2
Measure: Number; unit: Subjects
Arm/Group | Tritanrix-HepB/Hib-MenAC +Mencevax ACWY Group | Tritanrix-HepB/Hiberix+Mencevax ACWY Group
Number analyzed (Participants) | 192 | 69
Subjects
  anti-PSA ≥ 0.3 µg/mL (M24-30): number analyzed (Participants) | 182 | 66
  anti-PSA ≥ 0.3 µg/mL (M24-30) | 105 | 12
  anti-PSA ≥ 0.3 µg/mL (M25-31): number analyzed (Participants) | 192 | 68
  anti-PSA ≥ 0.3 µg/mL (M25-31) | 192 | 68
  anti-PSA ≥ 2 µg/mL (M24-30): number analyzed (Participants) | 182 | 66
  anti-PSA ≥ 2 µg/mL (M24-30) | 19 | 1
  anti-PSA ≥ 2 µg/mL (M25-31): number analyzed (Participants) | 192 | 68
  anti-PSA ≥ 2 µg/mL (M25-31) | 188 | 55
  anti-PSC ≥ 0.3 µg/mL (M24-30): number analyzed (Participants) | 191 | 69
  anti-PSC ≥ 0.3 µg/mL (M24-30) | 165 | 5
  anti-PSC ≥ 0.3 µg/mL (M25-31) | 192 | 69
  anti-PSC ≥ 2 µg/mL (M24-30): number analyzed (Participants) | 191 | 69
  anti-PSC ≥ 2 µg/mL (M24-30) | 23 | 0
  anti-PSC ≥ 2 µg/mL (M25-31) | 192 | 67

5. Secondary Outcome: Anti-PSA, Anti-PSC Antibody Concentrations
Description: Antibody concentrations were expressed as Geometric Mean Concentrations (GMCs).
Time Frame: Prior to (at 24 to 30 months of age) and after (at 25 to 31 months of age) Mencevax ACWY vaccination.
Population: as for outcome 2
Measure: Geometric Mean (95% Confidence Interval); unit: µg/mL
Arm/Group | Tritanrix-HepB/Hib-MenAC +Mencevax ACWY Group | Tritanrix-HepB/Hiberix+Mencevax ACWY Group
Number analyzed (Participants) | 192 | 69
µg/mL
  anti-PSA (M24-30): number analyzed (Participants) | 182 | 66
  anti-PSA (M24-30) | 0.42 [0.36 to 0.49] | 0.20 [0.17 to 0.24]
  anti-PSA (M25-31): number analyzed (Participants) | 192 | 68
  anti-PSA (M25-31) | 32.54 [27.79 to 38.10] | 6.94 [4.96 to 9.71]
  anti-PSC (M24-30): number analyzed (Participants) | 191 | 69
  anti-PSC (M24-30) | 0.72 [0.64 to 0.82] | 0.17 [0.15 to 0.19]
  anti-PSC (M25-31) | 35.13 [31.55 to 39.11] | 20.83 [16.60 to 26.15]

6. Secondary Outcome: Number of Subjects With Anti-hepatitis B Surface (Anti-HBs) Antigen Antibody Concentrations ≥ Cut-offs
Description: The antibody concentrations cut-off was ≥ 10 milli international units per millilitre (mIU/mL).
Time Frame: Prior to the Mencevax ACWY vaccination at 24-30 Months of age
Population: as for outcome 2
Measure: Number; unit: Subjects
Arm/Group | Tritanrix-HepB/Hib-MenAC +Mencevax ACWY Group | Tritanrix-HepB/Hiberix+Mencevax ACWY Group
Number analyzed (Participants) | 174 | 66
Subjects | 164 | 59

7. Secondary Outcome: Anti-HBs Concentrations
Description: Antibody concnetrations were expressed as Geometric Mean Concentrations (GMCs).
Time Frame: Prior to the Mencevax ACWY vaccination at 24-30 Months of age
Population: as for outcome 2
Measure: Geometric Mean (95% Confidence Interval); unit: mIU/mL
Arm/Group | Tritanrix-HepB/Hib-MenAC +Mencevax ACWY Group | Tritanrix-HepB/Hiberix+Mencevax ACWY Group
Number analyzed (Participants) | 174 | 66
mIU/mL | 251.1 [185.0 to 340.7] | 279.6 [162.5 to 481.0]

8. Secondary Outcome: Number of Subjects With Vaccine Response for rSBA-Men A, C
Description: Vaccine response was defined as follows: for initially seronegative subjects (i.e. with rSBA titer < 1:8 pre-vaccination), rSBA titer ≥ 1:32 post-vaccination (seroconversion), and for initially seropositive subjects (i.e. with rSBA > 1:8 prevaccination), at least a 4-fold increase in rSBA titer from pre-vaccination to post-vaccination.
Time Frame: 1 month after Mencevax ACWY vaccination (at 25 to 31 months of age).
Population: as for outcome 2
Measure: Number; unit: Subjects
Arm/Group | Tritanrix-HepB/Hib-MenAC +Mencevax ACWY Group | Tritanrix-HepB/Hiberix+Mencevax ACWY Group
Number analyzed (Participants) | 180 | 61
Subjects
  rSBA-MenA, Total: number analyzed (Participants) | 101 | 58
  rSBA-MenA, Total | 42 | 26
  rSBA-MenC, Total | 175 | 44

9. Secondary Outcome: Number of Subjects With Solicited Local Symptoms
Description: Assessed solicited local symptoms were pain, redness, swelling. Any = symptom occurring regardless of intensity grade.
Time Frame: During the 4-day follow-up period after the Mencevax ACWY vaccination, at 24-30 months of age
Population: The analysis were performed on the Booster Total Vaccinated Cohort included all subjects vaccinated during study NCT00291343.
Measure: Number; unit: Subjects
Arm/Group | Tritanrix-HepB/Hib-MenAC +Mencevax ACWY Group | Tritanrix-HepB/Hiberix+Mencevax ACWY Group
Number analyzed (Participants) | 203 | 93
Subjects
  Any Pain | 58 | 34
  Any Redness | 78 | 38
  Any Swelling | 48 | 28

10. Secondary Outcome: Number of Subjects With Solicited General Symptoms
Description: Assessed solicited general symptoms were drowsiness, irritability, loss of appetite, rectal fever [≥ 38 degrees Celsius (°C)]. Any = occurrence of symptom regardless of intensity grade.
Time Frame: During the 4-day follow-up period after the Mencevax ACWY vaccination, at 24-30 months of age
Population: as for outcome 9
Measure: Number; unit: Subjects
Arm/Group | Tritanrix-HepB/Hib-MenAC +Mencevax ACWY Group | Tritanrix-HepB/Hiberix+Mencevax ACWY Group
Number analyzed (Participants) | 203 | 93
Subjects
  Any Drowsiness | 23 | 7
  Any Irritability | 32 | 13
  Any Loss of appetite | 20 | 13
  Any fever (rectal) | 38 | 15

11. Secondary Outcome: Number of Subjects With Unsolicited Adverse Events (AEs)
Description: An unsolicited AE covers any untoward medical occurrence in a clinical investigation subject temporally associated with the use of a medicinal product, whether or not considered related to the medicinal product and reported in addition to those solicited during the clinical study and any solicited symptom with onset outside the specified period of follow-up for solicited symptoms. Any is defined as the occurrence of any unsolicited AE regard-less of intensity grade or relation to vaccination.
Time Frame: From Day 0 at months 15-24 of age to study end at Months 25-31 of age
Population: as for outcome 9
Measure: Number; unit: Subjects
Arm/Group | Tritanrix-HepB/Hib-MenAC +Mencevax ACWY Group | Tritanrix-HepB/Hiberix+Mencevax ACWY Group
Number analyzed (Participants) | 203 | 93
Subjects | 10 | 9

12. Secondary Outcome: Number of Subjects With Serious Adverse Events (SAEs)
Description: SAEs assessed include medical occurrences that result in death, are life threatening, require hospitalization or prolongation of hospitalization or result in disability/incapacity.
Time Frame: From 15-24 Months of age up to Months 25-31 of age
Population: as for outcome 9
Measure: Number; unit: Subjects
Arm/Group | Tritanrix-HepB/Hib-MenAC +Mencevax ACWY Group | Tritanrix-HepB/Hiberix+Mencevax ACWY Group
Number analyzed (Participants) | 203 | 93
Subjects | 6 | 1

ADVERSE EVENTS:
Time Frame: SAE(s): From Day 0 at Months 15-24 of age and up to study end at Months 25-31 of age. Solicited local/general symptoms: During the 4-day follow-up period after vaccination.
Arm/Group | Tritanrix-HepB/Hib-MenAC +Mencevax ACWY Group | Tritanrix-HepB/Hiberix+Mencevax ACWY Group
Serious Adverse Events (participants affected / at risk) | 6/203 | 1/93
Other Adverse Events (participants affected / at risk) | 125/203 | 59/93
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Tritanrix-HepB/Hib-MenAC +Mencevax ACWY Group (N=203) | Tritanrix-HepB/Hiberix+Mencevax ACWY Group (N=93)
Febrile convulsion (Nervous system disorders) | 1 | 0
Diarrhoea infectious (Infections and infestations) | 2 | 0
Gastroenteritis (Infections and infestations) | 1 | 0
Pulmonary tuberculosis (Infections and infestations) | 1 | 0
Urinary tract infection (Infections and infestations) | 1 | 0
Food intolerance (Metabolism and nutrition disorders) | 1 | 0
Amoebiasis (Infections and infestations) | 1 | 0
Ascariasis (Infections and infestations) | 1 | 0
Convulsion (Nervous system disorders) | 1 | 0
Electrolyte imbalance (Metabolism and nutrition disorders) | 1 | 0
Excoriation (Injury, poisoning and procedural complications) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Tritanrix-HepB/Hib-MenAC +Mencevax ACWY Group (N=203) | Tritanrix-HepB/Hiberix+Mencevax ACWY Group (N=93)
Pain (General disorders) | 58 | 34
Redness (General disorders) | 78 | 38
Swelling (General disorders) | 48 | 28
DROWSINESS (General disorders) | 23 | 7
IRRITABILITY (General disorders) | 32 | 13
LOSS OF APPETITE (General disorders) | 20 | 13
FEVER (General disorders) | 38 | 15

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.